CLINICAL TRIAL: NCT01067547
Title: A Randomised Controlled Trial Comparing the Efficacy of Intravenous Iron Sucrose and Oral Iron Sulfate in Patients With Iron Deficiency.
Brief Title: A Trial of Iron Replacement in Patients With Iron Deficiency.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Richard Fedorak (Other)
Responsible Party: Sponsor-Investigator, Richard Fedorak, Professor, Gastroenterology, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UA 2009 TL
Record Dates: First submitted 2009-11-12; First posted 2010-02-11 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Iron Deficiency; Inflammatory Bowel Disease
Keywords: Iron deficiency; Inflammatory Bowel Disease; Crohn's Disease; Ulcerative colitis
MeSH Terms: conditions — Iron Deficiencies; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iron sulfate (Experimental): Oral iron sulfate 300mg tid
  Interventions: Drug: Iron Sucrose.
- intravenous iron sulfate (Active Comparator): intravenous iron sulfate 300 mg
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron Sucrose. — The total dose of iron sucrose given will be individualised by calculating their iron deficit.
  Other Names: Iron sucrose is been marketed in Canada as Venofer.
  Arms: iron sulfate
Drug: Iron sucrose — 300mg of iron sucrose is given intravenously. Three infusions, each one week apart is given to patients with iron deficiency without anemia. For those patient with anemia, four infusions would be given.
  Other Names: Venofer
  Arms: intravenous iron sulfate

SUMMARY:
Primary Hypothesis: There is no difference in the efficacy of iron replacement by oral or intravenous route in Inflammatory Bowel Disease patients.

Iron deficiency anaemia is a common problem in people with inflammatory bowel disease (IBD) and patients with excessive blood loss from the bowel or heavy menstrual loss. Treatment options include a blood transfusion, oral iron with (Ferrograd ®) or intravenous iron replacement with iron sucrose (Venofer®). Iron deficiency anaemia is associated with poor quality of life, poor concentration span and low energy level. Blood transfusion may improve symptomatic anaemia quickly but there is a risk of transfusion reaction and blood born infection transmission. Moreover, packed cells are scarce resource therefore its use needs to be carefully prioritized. Oral iron supplement has been widely used and it can be purchased over the counter, however, its efficacy is not known in IBD population. Oral iron is poorly tolerated with side effects include altered bowel habit, nausea and darken stools, making it difficult to adhere to. In contrast, intravenous iron therapy with Venofer® has been shown to replenish iron store and improve anaemia quickly. To date, the safety of Venofer® use has been supported by its post marketing surveillance. Limitations with intravenous iron replacement include the need for medical supervision in the setting of limited healthcare resources; the need for patients to take multiple days off work and the cost of Venofer®. Currently it is uncertain which method of iron replacement is better. The purpose of this study is to compare the efficacy and the cost of oral and intravenous iron replacement in the setting of iron deficiency anaemia.

DETAILED DESCRIPTION:
1.1 Literature

Iron deficiency anemia is a common and a major management issue in Inflammatory Bowel disease [1-3]. Moreover, no factor has been identified in predicting recurrent iron deficiency anemia [4]. Iron deficiency and anemia are well recognized causes of fatigue, poor concentration and decreased energy level which impact on one's quality of life and ability to maintain employment or managing activities of daily living [2, 5]. Iron deficiency anemia is multi-factorial in origin and its causes can be divided into disease or patient origin. Disease factors include active blood loss from gastrointestinal mucosal ulceration, impairment of iron absorption if disease affects the proximal small bowels or a history of extensive small bowel resection. Iron absorption and utilization may also be influenced by inflammation inducible production of the hepatic origin peptide hormone called hepcidin [5], Interleukin 10 (IL10) [6] and interleukin 6 (IL 6) [7, 8]. Inflammatory cytokines such as Tumour Necrosis Factor alpha (TNFa) and IL-6 have been shown to cause anorexia in the animal model [9]. The major patient factor is dietary aversion of certain food in order to avoid exacerbation of existing symptom [10, 11].

Iron can be replaced either orally or intravenously. To date five studies directly compare oral versus intravenous iron therapy in patients with inflammatory bowel disease. Three of the studies suggested intravenous iron was superior [12-14], one suggested oral iron was superior [15]and one showed no difference[16]. This confusion is evident by a retrospective review of a gastroenterology outpatient clinic's experience in detecting and managing iron deficiency anaemia in both IBD and non IBD patients[17]. Furthermore, there are studies advocating the concurrent use of Erythropoietin which makes it difficult to draw a definite conclusion.

Studies have shown that iron deficient without anaemia is associated with reduced cognitive performance and it is reversible with iron supplementation.(18)19) In combination with other non specific symptoms such as fatigue and poor concentration span, many clinicians have been treating iron deficiency before anaemia occurs. Moreover, the World Health Organization (WHO) estimated the number of iron deficient people to be twice that of diagnosed anaemic people, (20) therefore, it is more appropriate to use iron deficiency as the inclusion criterion. This is in contrast with most of the clinical trials examining iron replacement therapy use iron deficiency anaemia as the inclusion criteria. The approach of stratifying the route of iron replacement therapy by the degree of anaemia is logical but not evidence based. This study seeks to investigate the efficacy of intravenous iron versus oral iron replacement in iron deficient patients.

Bone marrow biopsy staining for iron store is the gold standard for assessing iron store but it is invasive, therefore surrogate serum markers such as ferritin and iron saturation are used in clinical practice and they have been shown to be accurate.(21) Low ferritin level is associated with high (78%-100%) specificity and low iron saturation has a high sensitivity for iron deficiency (59%-88%). (22) Moreover, in anaemic IBD population, low ferritin level has >90% specificity for iron deficiency. (23) Given some of the IBD patients will have 'functional' iron deficiency with elevated ferritin and CRP and a low iron saturation, we have decided to use iron saturation <16% and ferritin less than 100ug/L to indicate iron deficient state. This cut off is consistent with the laboratory standard for University of Alberta Hospital.

1.2 Oral Iron Therapy

1.2.1 Oral Iron Adverse Events

Oral iron replacement is often poorly tolerated as evident by published studies where the adverse reaction rate has been reported to be as high as 80% [12], the discontinuation rate of up to 25% [16, 18]. Less than half of the patients were able to tolerate the prescribed dose of oral iron [14]. Some reports suggested oral iron therapy is associated with worsening of IBD disease activity [12], although not consistently [14]. Finally, there is controversy regarding whether or not oral iron replacement could exacerbate underlying disease through increased oxidative stress [18].

1.2.2. Oral Iron Efficacy

Semrin et al have demonstrated oral iron absorption is significantly impaired in the context of active Crohn's disease when compared to inactive disease state [7]. In the literature, the efficacy of oral iron replacement is often defined by an improvement in haemoglobin level by 20g/L or more from baseline and it has been reported to be as high as 89% [15]. It is worth noting that the baseline haemoglobin in the oral replacement cohort of the study by Gisbert et al was significantly higher than the intravenous cohort. When using iron studies as an endpoint, only 60% of oral iron treatment group were not iron deficient after 5 months of as tolerated dose of oral iron replacement [14].

1.3 Intravenous Iron Therapy

1.3.1 Intravenous Iron Adverse Events

The alternative to oral iron is intravenous iron replacement and its formulation has changed over time. Chertow et al reviewed the US FDA intravenous iron adverse event data between 2001-2003 and confirmed a up to 20 times higher rate of life threatening adverse events with the high molecular weight iron dextran than iron sucrose [19]. Iron sucrose (1.4+/- 0.5g) has been shown to increase HB by 20g/L and/or normalizing haemoglobin in up to 91% of the cohort within 12 weeks of treatment [20]. Studies have shown intravenous iron therapy is better tolerated than oral iron, with a lower discontinuation rate [13] and a definite improvement in the serum ferritin [16]. Intravenous iron replacement ensures adequate total iron replacement because there isn't an issue with compliance and it is independent from intestinal absorption. Iron sucrose has been shown to be efficacious when oral iron replacement is inadequate or intolerable [20]. The disadvantages of intravenous iron include it being time consuming for the patient, much more expensive than the oral formulation and the ancillary cost. It is uncertain what the true cost of intravenous iron replacement is without factoring in efficacy, compliance and the lack of side effect. Intravenous iron usage has been shown to be cost effective in chronic renal failure patients on dialysis who has insufficient iron stores on maximum tolerated oral supplements [21].

1.3.2 Intravenous Iron Efficacy

There have been five direct comparative oral versus intravenous iron replacement studies. The earlier comparative study involved smaller number of subjects, 19 patients, with short treatment duration of 2 weeks [12] and 6 weeks [16] and in one study, the baseline entry criterion between the two groups were different [15]. Appendix one summarises these studies.

1.4 Potential Aggravating Effects of Iron Therapy on Inflammatory Bowel Disease.

The role of oral iron in causing intestinal oxidative stress and subsequently increase the risk of colorectal dysplasia is a controversial one. Lund et al used 18 healthy volunteers to demonstrate that unabsorbed dietary iron is associated with a 40% increase in stool free radicals formation and carcinogens production [22]. The hypothesis that dietary iron can serve as a catalyst in the formation of highly reactive radical via the Fenton reaction [23, 24] and thereby causing cellular damage [25] and contributing to carcinogenesis has been demonstrated in animal models [26, 27]. A more recent mice model by Seril et al demonstrated the superiority of an intraperitoneal iron supplementation in replenishing splenic iron store without an increase in colorectal dysplasia rate compared to mice fed oral iron supplements [28]. Interestingly, there are conflicting reports regarding the role of intravenous iron replacement and the increase in plasma oxidative stress [12, 29] and the significance of this data is unknown. Currently, limited human literature is available addressing this issue.

HYPOTHESIS:

Primary:

There is no difference in the efficacy of iron replacement by oral or intravenous route in IBD patients.

Secondary:

There is no difference in the tolerability of oral and intravenous iron therapy.

The route of iron replacement does not impact on the colonic bacterial flora composition, the underlying IBD state and the oxidative stress of the colonic mucosa as determined by colonic biopsies analyzing for endoplasmic reticulum stress.

Oral iron replacement therapy is a cheap and efficacious way of replacing iron compare to intravenous replacement.

2 Trial Design

2.1 Primary Endpoint Change in iron saturation at week 8 post initiation of treatment.

2.2 Secondary Endpoints

To describe the change in haemoglobin, ferritin, IBDQ, HBI and partial MAYO score in patients before and after iron replacement.

To describe the changes in the colonic endoplasmic reticulum as an indicator of oxidative stress.

To describe the changes in urinary metabolomics from iron replacement To describe the change in the faecal bacteria composition pre and post iron replacement.

2.3 Study Design/Type

Open label Randomised Control Trial and observer blinded.

2.4 Randomization

Eligible all comers will be randomized into either IV or PO iron therapy in a 1:1 ratio.

Randomization will be performed externally and hold by EPICORE centre. EPICORE centre will maintain the randomization code.

3.1 Trial Treatment/ Duration

3.2 Dose determination:-

Total amount of intravenous iron given is calculated by Ganzoni Equation:

Iron dose (mg) = body weight (kg) x (ideal Hb - actual Hb) x 0.24 + 15mg/kg of iron depot

3.3 Iron Sucrose: Administered by IV infusion (dilute 5 mL (equiv. Fe 100 mg) in 100ml of NaCl 0.9%). Maximum amount of iron sucrose is 300mg per infusion per week.

3.4 Oral iron: 200mg equivalent of elemental iron is given twice a day for 3 months.

3.5 Discontinuation if

* withdrawal of consent
* Significant adverse event such as hypersensitivity reaction, dyspnoea and myalgia with iron sucrose. (see appendix 2)
* Recurrent intolerable non hypersensitivity reaction such as fatigue and GI disturbance.

3.6 Product Accountability Iron tablet pill count will take place during the monthly review.

3.7 Data Identification Appendix 3: Trial activity Schedule.

ELIGIBILITY:
Inclusion Criteria:

IBD group:

* Inflammatory Bowel Disease diagnosed by standard clinical, endoscopic and histological criteria
* Iron deficiency: Ferritin <12 if normal CRP or Ferritin <100 if elevated CRP AND/OR iron saturation < 16%
* stable dose of thiopurine or methotrexate for 1 month

Control group:

* Iron deficiency without IBD/ Coeliac disease/ haematological malignancy
* iron deficiency: Ferritin <12 if normal CRP or CRP <100 if elevated CRP AND/OR iron saturation < 16%

Exclusion Criteria:

Patients:

* with severe IBD who is likely to need hospitalization within 4 weeks of enrollment
* with untreated concurrent Vitamin B12 or folate deficiency at baseline
* with Coeliac disease
* pregnant and/or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Improvement of iron saturation at week 8. | month 0,2,3.

SECONDARY OUTCOMES:
To describe the change in the faecal bacteria composition pre and post iron replacement. | Three measurments - at month 0,3.
To describe the changes in ferritin, haemoglobin, Hepcidin,IBDQ, Modified HBI and partial MAYO score in patients before and after iron replacement. | month 0,2,3
To describe the changes in the colonic mucosal endoplasmic reticulum as an indicator of oxidative stress. | month 0 and 3.
To describe the changes in urinary metabolomics from iron replacement. | month 0,3.
Compare the health economics of intravenous versus oral iron replacement. | End of study.

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Fedorak, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Lee T, Clavel T, Smirnov K, Schmidt A, Lagkouvardos I, Walker A, Lucio M, Michalke B, Schmitt-Kopplin P, Fedorak R, Haller D. Oral versus intravenous iron replacement therapy distinctly alters the gut microbiota and metabolome in patients with IBD. Gut. 2017 May;66(5):863-871. doi: 10.1136/gutjnl-2015-309940. Epub 2016 Feb 4. PMID 26848182